CLINICAL TRIAL: NCT03012334
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, 5-Period, Cross-Over Study Assessing the Effects of Lasmiditan on Simulated Driving Performance in Normal Healthy Volunteers
Brief Title: The Effects of Lasmiditan on Simulated Driving Performance - Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Algorithme Pharma Inc (Industry); Cognitive Research Corporation (Industry); CoLucid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 16883; COL MIG-106 (Other: CoLucid Pharmaceuticals); H8H-CD-LAHG (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-12-27; First posted 2017-01-06 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lasmiditan 50mg (milligrams) (Experimental): Participants received 50mg of Lasmiditan tablets given as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
  Interventions: Drug: Lasmiditan
- Lasmiditan 100mg (Experimental): Participants received 100mg of Lasmiditan tablets given as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
  Interventions: Drug: Lasmiditan
- Lasmiditan 200mg (Experimental): Participants received 200mg of Lasmiditan tablets given as single doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
  Interventions: Drug: Lasmiditan
- Alprazolam 1mg (Active Comparator): Participants received 1mg of Alprazolam tablets as single oral dose on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
  Interventions: Drug: Alprazolam
- Placebo (Placebo Comparator): Participants received placebo tablets identical to Lasmiditan, administered as single oral dose on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Dose is based on treatment sequence in 5-way crossover
  Other Names: LY573144
  Arms: Lasmiditan 100mg; Lasmiditan 200mg; Lasmiditan 50mg (milligrams)
Drug: Alprazolam — Active comparator based on treatment sequence in 5-way crossover
  Arms: Alprazolam 1mg
Other: Placebo — Placebo comparator based on treatment sequence in 5-way crossover
  Arms: Placebo

SUMMARY:
This will be a randomized, single dose, double-blind, placebo-controlled, Latin-square design with 5-period (full) crossover study with participants randomized to treatment sequences. Participants will complete all 5 Periods.

During each Period, participants will come to the clinical research unit (CRU) and remain overnight before being dosed with a single dose of either lasmiditan, alprazolam, or placebo in the morning. Cognitive testing and driving simulation will be conducted post dosing. Participants will have a washout of at least 5 days between each Period.

This study is designed to test non-inferiority of lasmiditan doses relative to placebo, with an alprazolam test versus placebo to confirm the sensitivity of the simulator to detect treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to voluntarily consent to participate in this study and provide written informed consent prior to start of any study-specific procedures.
* Males and females between the ages of 21 and 50 years of age (inclusive). No more than 60% of one gender will be enrolled in the study.
* Body Mass Index (BMI) between 18 and 32 kilograms per meter squared (kg/m²) (inclusive).
* Participant is able to reliably perform study assessments (Standard Deviation of Lateral Position (SDLP) no higher than 1 standard deviation greater than the mean for normal healthy adults completing the practice scenario; Symbol Digit Coding (SDC) Correct no less than 1 standard deviation below the mean for healthy adults in their age range); demonstrates the ability to understand task instructions, and is physically capable (e.g., adequate manual dexterity, vision, and hearing) and cognitively capable of performing study tasks.
* Participant possesses a valid driver's license and is an active driver. Drives a minimum of 10,000 miles (about 16,000 km) per year for the previous 3 years.
* Participant must also demonstrate simulator sickness questionnaire scores which are not indicative of simulator sickness as defined in the driving simulation operations manual.
* Participant has a regular sleep pattern, is not engaged in shift-work, and in general, has at least 7 hours of sleep each night (bedtime occurs between 21:00 and 24:00 hours).
* Participant has a score < 10 on the Epworth Sleepiness Scale.
* Use of a medically highly effective form of birth control during the study and for thirty (30) days:
* Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* History or presence of clinically significant condition that, in the opinion of the Investigator, would jeopardize the safety of the participant or the validity of the study results.
* A history within 2 years of, or current treatment for, a sleeping disorder (including excessive snoring, obstructive sleep apnea), or a chronic painful condition that interferes with the participant's sleep.
* A history of difficulty either falling asleep or staying asleep in the previous 3 months, that is considered clinically significant by the investigator.
* Participant has a history or diagnosis of any of the following conditions:

  * Primary or secondary insomnia
  * Narcolepsy
  * Cataplexy (familial or idiopathic)
  * Circadian Rhythm Sleep Disorder
  * Parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and rapid eye movement behavior disorder
  * Sleep-related Breathing Disorder (obstructive or central sleep apnea syndrome, central alveolar hypoventilation syndrome)
  * Periodic Limb Movement Disorder
  * Restless Legs Syndrome
  * Primary Hypersomnia
  * Excessive Daytime Sleepiness (EDS)
  * Participant has visual or auditory impairment which in the opinion of the investigator would interfere with study related procedures or study conduct.
* Expected to use any other medication or dietary supplement to promote sleep including over- the-counter sleep medications, during their participation in the study.
* Participant consumes excessive amounts of coffee, tea, cola, or other caffeinated beverages per day.
* Participant has traveled across 1 or more time zones (transmeridian travel) in the last 2 weeks prior to randomization or is expected to travel across 1 or more time zones during the study.
* Expected to work on a rotating shift during their participation in the study.
* Participant works a night shift.
* History or presence of seizure disorder.
* History of urinary retention, angle closure glaucoma, or increased ocular pressure.
* History of gastrointestinal tract surgery, except for appendectomy.
* Has abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at Screening, that are considered clinically significant by the investigator.
* Presence of out-of-range cardiac interval on the screening ECG or other clinically significant ECG abnormalities
* History of orthostatic hypotension, fainting spells, or blackouts, that are considered clinically significant by the investigator.
* The presence of chronic or acute infections, that are considered clinically significant by the investigator.
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the study as judged by the Investigator.
* Use of psychoactive prescription or non-prescription medications, psychoactive nutritional supplements or herbal preparations within 2 weeks or 5 half-lives (whichever is longer) of admission to the clinical research unit (CRU) on Day -1.
* Has received any previous study drug within 30 days prior to the first dose of this study drug.
* Is a smoker of more than 10 cigarettes or eCigarettes, or 3 cigars or 3 pipes per day, and is unable to refrain from smoking while confined to the CRU.
* Has any history of dependency or treatment for substance abuse within the past 2 years.
* Participant with a history of alcoholism or who consumes excessive amounts of alcohol.
* Participants who consume alcohol on a regular basis (i.e., ≥ 5 times/week) before bedtime will be excluded from the study.
* Inability to comply with the dietary regimen of the clinical research center.
* Pregnancy / positive pregnancy test.
* Planning to become pregnant during the study or within 1 month of study completion.
* Inability to use adequate contraception during the study. It is recommended that adequate contraception be used for 30 days following completion of the study.
* Has a positive screen for alcohol or other drugs of abuse (amphetamines, methamphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has a history for Hepatitis B, Hepatitis C , or Human Immunodeficiency Virus (HIV) at Screening or has been previously treated for Hepatitis B, Hepatitis C, or HIV.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Algorithme Pharma, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with five study periods, each participant received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and Placebo as per the dosing sequence in each period. The washout period between dosing in consecutive study periods was at least 7 days.
Groups:
- Sequence 1: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 50 mg, Period 2: Lasmiditan 100 mg, Period 3: Placebo, Period 4: Lasmiditan 200 mg and Period 5: Alprazolam 1 mg
- Sequence 2: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 100 mg, Period 2: Lasmiditan 200 mg, Period 3: Lasmiditan 50 mg, Period 4: Alprazolam 1 mg and Period 5: Placebo
- Sequence 3: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 200 mg, Period 2: Alprazolam 1 mg, Period 3: Lasmiditan 100 mg, Period 4: Placebo and Period 5: Lasmiditan 50 mg
- Sequence 4: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Alprazolam 1 mg, Period 2: Placebo, Period 3: Lasmiditan 200 mg, Period 4: Lasmiditan 50 mg and Period 5: Lasmiditan 100 mg
- Sequence 5: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Placebo, Period 2: Lasmiditan 50 mg, Period 3: Alprazolam 1 mg, Period 4: Lasmiditan 100 mg and Period 5: Lasmiditan 200 mg
- Sequence 6: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Alprazolam 1 mg, Period 2: Lasmiditan 200 mg, Period 3: Placebo, Period 4: Lasmiditan 100 mg and Period 5: Lasmiditan 50 mg
- Sequence 7: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Placebo, Period 2: Alprazolam 1 mg, Period 3: Lasmiditan 50 mg, Period 4: Lasmiditan 200 mg and Period 5: Lasmiditan 100 mg
- Sequence 8: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 50 mg, Period 2: Placebo, Period 3: Lasmiditan 100 mg, Period 4: Alprazolam 1 mg and Period 5: Lasmiditan 200 mg
- Sequence 9: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 100 mg, Period 2: Lasmiditan 50 mg, Period 3: Lasmiditan 200 mg, Period 4: Placebo and Period 5: Alprazolam 1 mg
- Sequence 10: Participants received Lasmiditan (50 milligrams (mg), 100mg, and 200mg), Alprazolam 1mg and placebo as per the below dosing schedule.
  Period 1: Lasmiditan 200 mg, Period 2: Lasmiditan 100 mg, Period 3: Alprazolam 1 mg, Period 4: Lasmiditan 50 mg and Period 5: Placebo
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 8
Completed | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 8 | 9 | 8
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 8 | 9 | 8
Completed | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 8 | 9 | 8
Completed | 9 | 8 | 8 | 9 | 9 | 9 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 9 | 8 | 8 | 9 | 9 | 9 | 8 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 9 | 9 | 9 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 6 | 5 | 6 | 4 | 2 | 4 | 7 | 46
  Male | 6 | 5 | 4 | 3 | 4 | 3 | 5 | 7 | 5 | 2 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 3 | 2 | 3 | 2 | 0 | 0 | 0 | 15
  Not Hispanic or Latino | 7 | 7 | 8 | 6 | 7 | 6 | 7 | 9 | 9 | 9 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  White | 8 | 9 | 8 | 8 | 8 | 9 | 9 | 8 | 9 | 8 | 84
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 90

OUTCOME MEASURES:

1. Primary Outcome: Simulated Driving Performance in Healthy Participants as Measured by Standard Deviation of Lateral Position (SDLP) Using the Cognitive Research Corporation Driving Simulator-MiniSim (CRCDS-MiniSim)
Description: The standard deviation of lateral position (SDLP) is the primary parameter used as stable measure of driving performance with high test-retest reliability. It measures the driver's ability to stay in a constant position within the driving lane. Variations in the lateral position are recorded and analyzed. SDLP, was analyzed using a mixed model with fixed effects for sequence, period, and treatment, and a random effect for participant within sequence. A variance component covariance structure and Kenward-Roger degrees of freedom was used.
Time Frame: Approximately 90 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for simulated driving performance.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Groups:
- Lasmiditan 50mg: Participants received 50mg of Lasmiditan tablets given as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
- Lasmiditan 200mg: Participants received 200mg of Lasmiditan tablets given as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
- Alprazolam 1mg: Participants received 1mg of Alprazolam tablets as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Centimeters (cm) | 28.77 (6.73) | 38.52 (12.39) | 44.03 (13.55) | 50.24 (13.76) | 51.48 (14.47)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Non-Inferiority — Doses of lasmiditan were considered non-inferior to placebo if the upper 95% confidence limit on the difference in Standard Deviation of Lateral Position (SDLP) between that dose and placebo was less than 4.4 cm and lower doses also did not exceed the non-inferiority (NI) margin; p < .001, Mixed Models Analysis — P-value is obtained from mixed effect model for testing difference versus placebo equals to zero; LS Mean = 9.86, 95% CI 2-sided [7.39 to 12.33]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Non-Inferiority — Doses of lasmiditan were considered non-inferior to placebo if the upper 95% confidence limit on the difference in SDLP between that dose and placebo was less than 4.4 cm and lower doses also did not exceed the non-inferiority (NI) margin; p < 0.001, Mixed Models Analysis — P-value is obtained from mixed effect model for testing difference versus placebo equals to zero; LS Mean = 15.35, 95% CI 2-sided [12.87 to 17.82]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Mixed Models Analysis — P-value is obtained from mixed effect model for testing difference versus placebo equals to zero; LS Mean = 21.06, 95% CI 2-sided [18.60 to 23.52]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = 22.71, 95% CI 2-sided [20.23 to 25.18]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -12.85, 95% CI 2-sided [-15.32 to -10.38]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -7.36, 95% CI 2-sided [-9.84 to -4.88]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p = 0.19, Mixed Models Analysis; LS Mean = -1.65, 95% CI 2-sided [-4.11 to 0.82]

2. Secondary Outcome: Karolinska Sleepiness Scale (KSS) Score
Description: The KSS is used to assess subjective level of sleepiness. This is a participant self-report measure of situational sleepiness and provides an assessment of alertness/sleepiness at a particular point in time. It is a 9-point categorical Likert scale on which the participant rates sleepiness from 1 (very alert) to 9 (very sleepy/fighting sleep), with higher scores indicating more sleepiness and lower scores indicating more alertness.
Time Frame: Approximately 85 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for karolinska sleepiness scale.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Units on a scale | 2.8 (1.35) | 4.4 (1.85) | 5.1 (1.89) | 5.7 (1.94) | 6.2 (1.85)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 1.6, 95% CI 2-sided [1.1744 to 2.0335]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 2.3, 95% CI 2-sided [1.8306 to 2.6926]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 2.9, 95% CI 2-sided [2.4239 to 3.2800]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 3.4, 95% CI 2-sided [2.9568 to 3.8193]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -1.8, 95% CI 2-sided [-2.2137 to -1.3546]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -1.1, 95% CI 2-sided [-1.5574 to -0.6956]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p = 0.0142, Mixed Models Analysis; LS Mean = -0.5, 95% CI 2-sided [-0.9642 to -0.1081]

3. Secondary Outcome: Percentage of Participants With Self-Reported Readiness to Drive
Description: On each dosing day participants were asked "Right now do you feel safe to drive?". Pair-wise comparisons for readiness to drive were analyzed using McNemar test.
Time Frame: Approximately 85 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for self-reported readiness to drive.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Percentage of Participants | 100 | 80 | 67.9 | 55.3 | 43.5

4. Secondary Outcome: Motivational and Self-Appraisal Visual Analog Scale (VAS)
Description: After completing the driving simulation, participants assessed their own performance and their level of motivation to perform at their best during the driving simulation. Participants responded to 2 questions: 1. How well do you think you drove for the last 60 minutes? 2. How motivated did you feel to drive at your best during the last 60 minutes of driving?. Participants recorded their response to each question by writing a vertical line on a 100 millimeters (mm) horizontal, linear visual analog scale indicating their level of performance (Not Satisfactory to Satisfactory) and motivation (Not Motivated to Motivated). Scores on the 100 mm linear scale were measured to the nearest millimeter from the left. Scores ranged from 0-100 mm, with higher scores indicating motivated and satisfactory and lower scores indicating not motivated and not satisfactory.
Time Frame: Approximately 2.5 hours post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for visual analog scale.
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Millimeters (mm)
  VAS Motivation | 78.0 (18.48) | 65.6 (26.21) | 53.7 (30.98) | 49.9 (33.70) | 47.6 (33.86)
  VAS Self-appraisal | 77.2 (15.96) | 51.2 (27.03) | 39.8 (27.82) | 30.8 (25.17) | 24.7 (26.48)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -12.6, 95% CI 2-sided [-18.6895 to -6.5006]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -24.2, 95% CI 2-sided [-30.3631 to -18.1357]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -28.4, 95% CI 2-sided [-34.4420 to -22.2897]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -30.4, 95% CI 2-sided [-36.5068 to -24.2770]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 17.8, 95% CI 2-sided [11.7029 to 23.8908]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p = 0.0489, Mixed Models Analysis; LS Mean = 6.1, 95% CI 2-sided [0.0297 to 12.2554]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p = 0.5123, Mixed Models Analysis; LS Mean = 2.0, 95% CI 2-sided [-4.0500 to 8.1021]
Statistical Analysis 8: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -26.4, 95% CI 2-sided [-32.4956 to -20.3628]
Statistical Analysis 9: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -37.8, 95% CI 2-sided [-43.9270 to -31.7537]
Statistical Analysis 10: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -46.8, 95% CI 2-sided [-52.8147 to -40.7268]
Statistical Analysis 11: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -52.6, 95% CI 2-sided [-58.6490 to -46.4682]
Statistical Analysis 12: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 26.1, 95% CI 2-sided [20.0635 to 32.1953]
Statistical Analysis 13: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 14.7, 95% CI 2-sided [8.6325 to 20.8040]
Statistical Analysis 14: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p = 0.0605, Mixed Models Analysis; LS Mean = 5.8, 95% CI 2-sided [-0.2560 to 11.8317]

5. Secondary Outcome: Number of Correct Responses in Driving Performance Using CogScreen Symbol Digit Coding (SDC) Test
Description: The SDC Test, a digit symbol substitution test that is sensitive to changes in information processing speed, provides measures of response speed and accuracy. The test was administered prior to the simulated driving sessions. The principal test score measures the number of correct responses in 120 seconds. SDC was used in this study to measure attention, visual scanning, working memory, and speed of information processing. Scores range from 0 (No correct responses). A higher score indicates greater processing speed.
Time Frame: Approximately 85 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for driving performance.
Measure: Mean (Standard Deviation); unit: Responses
Groups:
- Alprazolam 1mg: Participants received 1mg Alprazolam tablets as single oral doses on Day 1, 7, 14, 21, or 28 (dependent upon the assigned treatment sequence) in the morning.
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Responses | 72.8 (10.18) | 68.1 (10.19) | 66.0 (8.78) | 64.1 (8.07) | 61.7 (10.10)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -4.5, 95% CI 2-sided [-6.14 to -2.85]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -6.9, 95% CI 2-sided [-8.58 to -5.28]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -8.9, 95% CI 2-sided [-10.52 to -7.23]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -11.2, 95% CI 2-sided [-12.81 to -9.51]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = 6.7, 95% CI 2-sided [5.02 to 8.31]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = 4.2, 95% CI 2-sided [2.58 to 5.88]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p < 0.007, Mixed Models Analysis; LS Mean = 2.3, 95% CI 2-sided [0.64 to 3.93]

6. Secondary Outcome: Driving Performance Using the CRCDS-MiniSim - Lane Exceedance
Description: The CRCDS-MiniSim is a PC-based research driving simulator that provides a realistic automotive driving environment. The present study employs the Country Vigilance-Divided Attention (CVDA) driving scenario, a 62.1 mile (100 km), monotonous, two lane highway driving task that includes a secondary visual vigilance task (DA). The monotonous Country Vigilance scenario has been demonstrated to be sensitive to detect the effects of fatigue or sleepiness on driving performance. Lane exceedance is the number of lane exceedances, an indication of lane position control, (i.e., the driver's ability to stay within his/her lane), as measured by the number of times that the front left or right tire of the vehicle crosses over the right or left lane boundary.
Time Frame: Approximately 90 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for driving performance.
Measure: Mean (Standard Deviation); unit: Lane Exceedances
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Lane Exceedances | 2.288 (1.3406) | 3.716 (1.3336) | 4.301 (1.1496) | 4.884 (0.8359) | 4.841 (0.8575)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 1.439, 95% CI 2-sided [1.2198 to 1.6583]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 2.018, 95% CI 2-sided [1.7981 to 2.2380]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 2.572, 95% CI 2-sided [2.3536 to 2.7909]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = 2.553, 95% CI 2-sided [2.3331 to 2.7730]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -1.114, 95% CI 2-sided [-1.3333 to -0.8948]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -0.535, 95% CI 2-sided [-0.7549 to -0.3151]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p = 0.8629, Mixed Models Analysis; LS Mean = 0.019, 95% CI 2-sided [-0.1995 to 0.2379]

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Data presented are the number of participants who experienced 1 or more AEs (all causalities and drug-related) and serious AEs (SAEs). A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Up To 35 days
Population: All randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
Participants
  Other AEs | 8 | 34 | 47 | 62 | 71
  SAEs | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Driving Performance Using the CRCDS-MiniSim - Speed Deviation
Description: The CRCDS-MiniSim is a PC-based research driving simulator that provides a realistic automotive driving environment. The present study employs the Country Vigilance-Divided Attention (CVDA) driving scenario, a 62.1 mile (100 km), monotonous, two lane highway driving task that includes a secondary visual vigilance task (DA). The monotonous Country Vigilance scenario has been demonstrated to be sensitive to detect the effects of fatigue or sleepiness on driving performance. Speed deviation is a measure of intra-individual variability. Measures that assess an individual's failure to maintain consistent performance are more sensitive to sedation than are measures of absolute performance.
Time Frame: Approximately 90 minutes post dose, on Day 1, 7, 14, 21, or 28 depending upon the assigned treatment sequence
Population: All randomized participants who received study drug and have evaluable data for driving performance.
Measure: Mean (Standard Deviation); unit: meter per second (m/sec)
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
Number analyzed (Participants) | 85 | 87 | 86 | 89 | 85
meter per second (m/sec) | 0.635 (0.2716) | 0.814 (0.3475) | 0.935 (0.5696) | 1.013 (0.4581) | 1.238 (0.5856)
Statistical Analysis 1: Comparison: Placebo vs Lasmiditan 50mg; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS Mean = 0.180, 95% CI 2-sided [0.0849 to 0.2746]
Statistical Analysis 2: Comparison: Placebo vs Lasmiditan 100mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 0.303, 95% CI 2-sided [0.2082 to 0.3985]
Statistical Analysis 3: Comparison: Placebo vs Lasmiditan 200mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 0.372, 95% CI 2-sided [0.2770 to 0.4662]
Statistical Analysis 4: Comparison: Placebo vs Alprazolam 1mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = 0.603, 95% CI 2-sided [0.5080 to 0.6983]
Statistical Analysis 5: Comparison: Lasmiditan 50mg vs Alprazolam 1mg; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean = -0.423, 95% CI 2-sided [-0.5183 to -0.3286]
Statistical Analysis 6: Comparison: Lasmiditan 100mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -0.300, 95% CI 2-sided [-0.3949 to -0.2047]
Statistical Analysis 7: Comparison: Lasmiditan 200mg vs Alprazolam 1mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean = -0.232, 95% CI 2-sided [-0.3261 to -0.1370]

ADVERSE EVENTS:
Time Frame: Up To 35 days
Description: All randomized participants who received study drug.
Arm/Group | Placebo | Lasmiditan 50mg | Lasmiditan 100mg | Lasmiditan 200mg | Alprazolam 1mg
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/87 | 0/86 | 0/89 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/85 | 0/87 | 0/86 | 0/89 | 0/85
Other Adverse Events (participants affected / at risk) | 8/85 | 34/87 | 47/86 | 62/89 | 71/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Lasmiditan 50mg (N=87) | Lasmiditan 100mg (N=86) | Lasmiditan 200mg (N=89) | Alprazolam 1mg (N=85)
Cerebellar haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Lasmiditan 50mg (N=87) | Lasmiditan 100mg (N=86) | Lasmiditan 200mg (N=89) | Alprazolam 1mg (N=85)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5) | 6 (6) | 3 (3)
Fatigue (General disorders) | 2 (2) | 15 (15) | 10 (11) | 7 (7) | 14 (14)
Dizziness (Nervous system disorders) | 1 (1) | 14 (14) | 18 (18) | 36 (37) | 26 (26)
Headache (Nervous system disorders) | 3 (3) | 8 (8) | 3 (3) | 5 (6) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4) | 7 (7) | 3 (3)
Somnolence (Nervous system disorders) | 2 (2) | 10 (10) | 23 (23) | 38 (38) | 45 (45)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and its results shall not be publicized in any form without prior consent of the Sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT03012334/SAP_000.pdf
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03012334/Prot_001.pdf